CLINICAL TRIAL: NCT00102856
Title: Neuromodulation and Language Acquisition (KS-Neuromod_01, Stage Ib)
Brief Title: Neuromodulation and Language Acquisition (Stage Ib)
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KS-NEUROMOD_01, Stage Ib; IZKF Muenster: Kne3/074/04
Record Dates: First submitted 2005-02-03; First posted 2005-02-04 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2006-09

CONDITIONS: Healthy
Keywords: language acquisition; plasticity; stroke recovery; associative learning
MeSH Terms: interventions — Pramipexole; Rivastigmine

INTERVENTIONS:
Drug: Pramipexole
Drug: Rivastigmine

SUMMARY:
The purpose of this study is to determine whether rivastigmine or pramipexol are effective in boosting semantic language acquisition in healthy subjects.

DETAILED DESCRIPTION:
Our prior work shows that d-amphetamine and the dopamine precursor levodopa markedly improve word learning success in healthy subjects. In this randomized, placebo-controlled, double-blind clinical trial, we probe whether a selective d2/d3 dopamine agonist (pramipexole) or cholinergic neuromodulation (rivastigmine), after a titration period of five days, will yield a learning enhancement comparable to using levodopa in healthy subjects. The expected scientific results will strengthen the basis for transferring neuromodulatory interventions from the laboratory to stroke patients with language dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* 20-35 years old
* Right handedness
* Left language dominance (as assessed by functional transcranial Doppler ultrasonography [fTCD])

Exclusion Criteria:

* Neurological/psychiatric/metabolic/cardiac disorders
* Asthma
* Known allergic reactions to one of the experimental drugs
* Other drugs affecting the central nervous system
* Leisure drug ingestion during the past 4 weeks (urine test)
* Smoking cessation during the past 2 weeks
* > 6 cups of coffee or energy drinks per day
* > 10 cigarettes per day
* > 50 grams of alcohol per day

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2005-01; Study Completion 2006-06

PRIMARY OUTCOMES:
Boost in language learning success (percent hits) through neuromodulation

SECONDARY OUTCOMES:
Stability of language learning success after one week, one month, and one year

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Breitenstein, PhD, Study Director — Dept. of Neurology, University Hospital Muenster; Stefan Knecht, MD, Study Chair — Dept. of Neurology, University Hospital Muenster
Locations (1):
- Dept. of Neurology, University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Knecht S, Breitenstein C, Bushuven S, Wailke S, Kamping S, Floel A, Zwitserlood P, Ringelstein EB. Levodopa: faster and better word learning in normal humans. Ann Neurol. 2004 Jul;56(1):20-6. doi: 10.1002/ana.20125. PMID 15236398
- [Background] Breitenstein C, Wailke S, Bushuven S, Kamping S, Zwitserlood P, Ringelstein EB, Knecht S. D-amphetamine boosts language learning independent of its cardiovascular and motor arousing effects. Neuropsychopharmacology. 2004 Sep;29(9):1704-14. doi: 10.1038/sj.npp.1300464. PMID 15114342